CLINICAL TRIAL: NCT06897917
Title: Real World Study of Oxycodone/Naloxone Sustained-Release Tablets (Mimeixin) for Patients With Severe Cancer Pain
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMX-RWS-01
Record Dates: First submitted 2025-03-05; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Opioid-Induced Constipation; Pain Cancer
Keywords: opioid-induced constipation; severe cancer pain; Oxycodone/naloxone sustained-release tablets
MeSH Terms: conditions — Opioid-Induced Constipation; Cancer Pain | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Oxycodone/naloxone sustained-release tablets treatment group (Experimental): Patients receiving oxycodone naloxone sustained-release tablets were included in the study cohort.
  Interventions: Drug: Oxycodone Hydrochloride and Naloxone Hydrochloride Sustained-release Tablets

INTERVENTIONS:
Drug: Oxycodone Hydrochloride and Naloxone Hydrochloride Sustained-release Tablets — 1. Calculate the total opioid dosage administered to the patient in the previous 24 hours and convert it to an equivalent dose of oxycodone/naloxone sustained-release tablets(Mimeixin).
  2. Based on the principle of incremental dosing, calculate the total dosage to be administered on the day of enrollment, divide it into two portions, and administer one portion every 12 hours (q12h).
  3. In case of breakthrough pain during treatment, administer an equivalent dose of immediate-release morphine or other medications equivalent to 10%-20% of the 24-hour background dosing for relief.
  4. If the number of breakthrough pain events exceeds 2 in a day after dosing, adjust the dosage again based on the incremental dosing principle. Adjustments should be made every 1-2 days, with each adjustment increasing the dose by a gradient of 5 mg/2.5 mg or 10 mg/5 mg of oxycodone/naloxone sustained-release tablets, twice daily, and so on. The maximum daily dose of oxycodone should not exceed 160 mg.
  Other Names: Mimeixin

SUMMARY:
This study is a prospective, single-arm, multicenter, real-world study to evaluate effect of bowel function, analgesic effect, quality of life, and safety of Mimeixin® in Chinese patients with severe cancer pain.

DETAILED DESCRIPTION:
Cancer remains a significant health concern globally, with rising incidence and mortality rates. In 2022, there were 19.96 million new cancer cases and 9.74 million cancer deaths worldwide, including 4.8 million new cases and 2.6 million deaths in China. Cancer patients often experience pain during treatment, with 40% of patients reporting persistent pain, particularly moderate to severe pain, occurring in 40%-80% of cases. Unrelieved pain can exacerbate symptoms such as anxiety, depression, fatigue, insomnia, and loss of appetite, significantly impacting patients' quality of life. Opioids, represented by morphine and oxycodone, are widely used for the treatment of moderate to severe cancer pain.

Long-term opioid use often leads to gastrointestinal adverse events, with opioid-induced constipation (OIC) being the most common, significantly affecting patients' quality of life and treatment compliance. Although some guidelines recommend laxatives as prophylactic and first-line treatment for OIC, approximately half of the patients do not experience adequate symptom improvement. The mechanism of OIC primarily involves the activation of intestinal μ-opioid receptors, which is difficult to address solely with laxatives. The key to treating OIC lies in blocking the stimulation of μ-opioid receptors in the gastrointestinal tract while maintaining the analgesic effect of opioid receptors in the central nervous system.

Oxycodone/naloxone sustained-release tablets, a combination of the opioid receptor agonist oxycodone and the antagonist naloxone, effectively provide analgesia while improving OIC. Foreign studies have demonstrated that this medication significantly improves OIC while maintaining good analgesic effects, with good long-term tolerability. Mimeixin® is an oxycodone/naloxone sustained-release tablet developed with reference to the foreign-listed drug Targin®. It was approved by the National Medical Products Administration of China in June 2024 for the treatment of severe pain in adults that requires opioid analgesics for adequate control. However, clinical validation has not been conducted among Chinese cancer pain patients. Therefore, a prospective, single-arm, multicenter, real-world study is planned to evaluate the effect in bowel function, analgesic effect, quality of life, and safety of Mimeixin® in Chinese patients with severe cancer pain in real-world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, with a histological or pathological diagnosis of advanced cancer.
* Be diagnosed with severe (NRS ≥ 7 points) cancer pain, requiring regular opioid therapy.
* Diagnosed with OIC according to the Rome IV diagnostic criteria for OIC, with a BFI score ≥ 30.
* Determined by the investigator to be eligible for treatment with oxycodone/naloxone sustained-release tablets.
* Estimated survival period of more than 3 months.
* Voluntarily sign an informed consent form.

Exclusion Criteria:

* Patients with contraindications to oxycodone/naloxone sustained-release tablets (including allergy to the active ingredients or any excipients of this product; severe respiratory depression accompanied by hypoxemia and/or hypercapnia; severe chronic obstructive pulmonary disease; pulmonary heart disease; severe bronchial asthma; paralytic ileus caused by non-opioid drugs; moderate to severe liver function impairment).
* Patients with structural malformations of the gastrointestinal tract (such as intestinal obstruction, stenosis), other known gastrointestinal diseases/symptoms (including cancer metastasis to the digestive tract), or gastrointestinal digestion and absorption disorders.
* Patients with language communication barriers, cognitive impairments or mental illnesses, intracranial metastasis of tumors with consciousness disorders, or consciousness disorders caused by other reasons.
* Other situations that the investigator judges as unsuitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes of Patients' Bowel Function of day 28 | pre-intervention, day 7, day 14, day 21 and day 28 after the intervention
  The BFI score was used for evaluation, and the data were repeatedly measured. A one-way repeated measures ANOVA model was used, which included follow-up time and baseline BFI values; the variation curve of BFI with follow-up time was also plotted. The analytical method for repeatedly measured data of secondary endpoints was consistent with the primary analytical method.

SECONDARY OUTCOMES:
Changes of Cancer Pain with NRS | through study completion, an average of 4 weeks
  Assess and record pain experienced within 24 hours using the Numerical Rating Scale (NRS) The numerical rating scale (NRS) uses 0-10 to represent different levels of pain, with higher scores indicating higher levels of pain.
Changes of Cancer Pain with BPI-SF | through study completion, an average of 4 weeks
  Assess and record pain experienced concurrently with the Brief Pain Inventory-Short Form (BPI-SF).
  The Brief Pain Inventory-Short Form (BPI-SF) was used to assess the degree of pain effect in the past 24 hours on a scale of 0-10, with 0 as no effect and 10 as complete effect.
Changes of breakthrough pain | within 24 hours
  Documented the frequency of breakthrough pain within 24 hours, as well as the types and amounts of rescue medications used within 24 hours.
Frequency of bowel movements and CSBMs | through study completion, an average of 4 weeks
  Documented the number of bowel movements and CSBMs.CSBM is defined as a spontaneous bowel movement accompanied by a complete sense of emptying, without the use of rescue laxatives or manual assistance.
Laxative Use | through study completion, an average of 4 weeks
  Record the type and amount of laxatives used.
Assessment of withdrawal symptoms | pre-intervention, day 2 and day 28 after the intervention
  Recorded using Subjective Opioid Withdrawal Scale (SOWS).
Changes of Quality of Life with EQ-5D-5L | day 7, day 14, day 21 and day 28 after the intervention
  The EQ-5D-5L consists of two main components: the EQ-5D Descriptive System and the EQ-5D Visual Analogue Scale (VAS). A score of 1-5 and a score of 0-100 were used to describe health status, with higher EQ-5D Descriptive System scores indicating worse health status and higher EQ-5D VAS scores indicating better health status.
Changes of Quality of Life with SF-6D | day 7, day 14, day 21 and day 28 after the intervention
  The SF-6D describes health status on a scale of 0-5. The best health status was "111111", and the worst health status was "555655".
Changes of Quality of Life with PAC-QOL | day 7, day 14, day 21 and day 28 after the intervention
  The PAC-QOL assesses the impact of constipation on your daily life over the past 2 weeks. It consists of 28 questions, each scored from 0 to 4.
Incidence of adverse events (Safety Evaluation) | through study completion, an average of 4 weeks
  The grading criteria for adverse events follow the Common Terminology Criteria for Adverse Events 5.0 (CTCAE 5.0) of the National Cancer Institute (NCI).

CONTACTS AND LOCATIONS:
Overall Officials: Suxia Luo, Doctor, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No